CLINICAL TRIAL: NCT01305447
Title: Getting Physical on Cigarettes: Exercise and Smoking Cessation - Preventing Relapse
Brief Title: Getting Physical on Cigarettes - Smoking Cessation & Relapse Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prapavessis NCIC RCT
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2012-06

CONDITIONS: Cancer
Keywords: smoking cessation; exercise maintenance; preventing relapse; weight gain; group-mediated cognitive behavioural therapy
MeSH Terms: conditions — Neoplasms; Smoking Cessation; Weight Gain | interventions — Exercise; Secondary Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise Maintenance (Experimental): Randomization and Group-Mediated Cognitive Behavioural therapy (GMCB) sessions will begin on week 8 of the program. Topics of self-regulation related to exercise (Social cognitive theory of self-regulation, Albert Bandura, 1991) will be discussed: monitoring, scheduling, goal setting, coping, overcoming barriers, rewards, social support.
  Following the termination of the 14 week exercise aided smoking cessation program, trained exercise facilitators will deliver 15 minute biweekly (for the first month), monthly (for the next 2 months), and then bimonthly (for last 8 months) intervention strategies over the phone to continue to enhance the GMCB principles on how to maintain exercise behavior.
  Interventions: Behavioral: Exercise Behaviour Maintenance
- Ex. Maintenance + relapse prevention (Experimental): The same topics of self-regulation related to exercise maintenance(Social cognitive theory of self-regulation, Albert Bandura, 1991) will be discussed: monitoring, scheduling, goal setting, coping, overcoming barriers, rewards, social support.
  Following the termination of the 14 week exercise aided smoking cessation program, trained exercise facilitators will deliver 15 minute biweekly (for the first month), monthly (for the next 2 months), and then bimonthly (for last 8 months) intervention strategies over the phone to continue to enhance the Group-Mediated Cognitive Behavioural therapy (GMCB) principles on how to maintain exercise behavior.
  Participants in this arm will also receive the Brandon et al. (2004) Forever Free smoking relapse prevention booklets.
  Interventions: Behavioral: Exercise Behaviour Maintenance; Behavioral: Smoking Relapse prevention booklets
- relapse prevention (Active Comparator): Randomization and group discussion sessions will begin on week 8 of the program. Topics of women's health, unrelated to exercise will be discussed (control).
  Following the termination of the 14 week exercise aided smoking cessation program, trained exercise facilitators will deliver 15 minute biweekly (for the first month), monthly (for the next 2 months), and then bimonthly (for last 8 months) phone calls to continue to maintain contact time.
  Participants in this arm will also receive the Brandon et al. (2004) Forever Free smoking relapse prevention booklets.
  Interventions: Behavioral: Smoking Relapse prevention booklets
- Contact Control (Active Comparator): Randomization and group discussion sessions will begin on week 8 of the program. Topics of women's health, unrelated to exercise will be discussed (control).
  Following the termination of the 14 week exercise aided smoking cessation program, trained exercise facilitators will deliver 15 minute biweekly (for the first month), monthly (for the next 2 months), and then bimonthly (for last 8 months) phone calls to continue to maintain contact time.
  Interventions: Behavioral: Contact control

INTERVENTIONS:
Behavioral: Exercise Behaviour Maintenance — Following the termination of the 14 week exercise aided smoking cessation program, trained exercise facilitators will deliver 15 minute biweekly (for the first month), monthly (for the next 2 months), and then bimonthly (for last 8 months) phone calls to remind the participants of the self-regulatory skills they learned during group discussion.
  Other Names: Physical Activity
  Arms: Ex. Maintenance + relapse prevention; Exercise Maintenance
Behavioral: Smoking Relapse prevention booklets — Participants will be given Brandon et al. (2000, 2004) smoking relapse prevention booklets following exercise program.
  Other Names: Educational material, relapse prevention, Forever Free
  Arms: Ex. Maintenance + relapse prevention; relapse prevention
Behavioral: Contact control — No treatment, but equal contact time as the other intervention arms. Topics of women's health, unrelated to exercise will be discussed in group-mediated sessions(control).
  Other Names: Control
  Arms: Contact Control

SUMMARY:
Adult female smokers will participate in an exercise-aided smoking cessation program, and will then be randomized into one of four cessation maintenance conditions: (a) Exercise Maintenance only (b) Exercise Maintenance + Relapse Prevention Booklets(c) Relapse Prevention Booklets + Contact and (d) Contact Control. Primary follow-up outcome is smoking behaviour. Secondary outcomes include exercise behaviour, Physiological measures (body composition (Dual-emission X-ray absorptiometry; DXA), vascular health (stiffness, endothelial function, carotid plaque volume), physical fitness), and Psychological measures (self-regulatory cognitions related to exercise adherence [exercise, scheduling, barrier, relapse, and concurrent self-regulatory self-efficacy]).

The hypotheses detailed below are specific to the randomization of participants into the following 4 groups:

1. Exercise Maintenance only
2. Exercise Maintenance + Relapse Prevention Booklets
3. Relapse Prevention Booklets + Contact
4. Contact Control

Hypothesis 1: Compared to quitters in the contact control condition, quitters exposed to a home-based lifestyle exercise maintenance intervention (Exercise Maintenance only and Exercise Maintenance + Relapse Prevention Booklets) will demonstrate significantly greater exercise adherence and fitness levels, as well as significantly less weight gain and smoking relapse rates following exercise-aided smoking cessation program termination.

Hypothesis 2: Compared to quitters in the contact control condition, quitters exposed to relapse information only (Relapse Prevention Booklets + Contact) will experience significantly less smoking relapse following exercise-aided smoking cessation program termination.

Due to the novelty and exploratory nature of the respective prevention programs, no hypotheses are specified with respect to which prevention program (exercise maintenance or relapse prevention information) will be superior to the other, or whether the additive benefits (i.e., exercise maintenance plus relapse prevention information) will be superior to one prevention program alone.

DETAILED DESCRIPTION:
Adding exercise to cognitive behaviour therapy (CBT) has been shown to aid smoking cessation and lessen some of the negative consequences of withdrawal symptoms (Marcus et al., 1999; Ussher, 2005). Recently, Prapavessis and colleagues (2007) demonstrated that their 12-week program, consisting of supervised vigorous intensity exercise as an adjunct to nicotine replacement therapy (NRT), facilitates smoking cessation, improves physical fitness, and delays weight gain in women smokers. However, a smoking relapse effect was shown post-intervention, illustrating a trend where, as abstinence decreased, physical fitness showed a corresponding decrease and an increase in weight (also see, Marcus et al.). These results suggest that exercise needs to be maintained if it is to be an effective aid to smoking cessation.

In practice, long-term supervised and structured vigorous exercise regimes are beyond the scope of smoking cessation services. Therefore, it is important to determine whether an exercise intervention program can be developed to maintain weight and physical fitness after program termination, and thus prevent (or reduce) smoking relapse. Teaching smokers the necessary self-regulatory skills needed to abstain from smoking and adhere to exercise independently may be a promising avenue through which to ensure lasting health behaviour changes.

The Getting Physical on Cigarettes program will begin in January 2010. The main purpose of this project is to examine whether an inexpensive, home-based lifestyle exercise maintenance intervention can demonstrate sustained health benefits in terms of weight gain and physical fitness benefits following an exercise and Nicotine Replacement Therapy (NRT) aided smoking cessation program. In addition, this trial seeks to examine previously unexplored topics of interest in the smoking abstinence literature; specifically, we are interested in whether the nicotine metabolite ratio (3-HC/Cotinine: Schnoll et al., 2009) is a useful biomarker for determining cessation success in relation to exercise and Nicotine Replacement Therapy (NRT) treatment, and whether the interactive effects of exercise and smoking cessation improve vascular health and lung function.

Four hundred and twenty adult female smokers will follow a structured and supervised 14 week exercise-aided smoking cessation program, with the 10 week NRT program beginning at week 4. Participants will be randomized into one of four conditions: a) Exercise Maintenance; b) Exercise Maintenance + Relapse Prevention Booklets; c) Relapse Prevention Booklets + Contact; and d) Contact Control. Starting at week 8, women in the Exercise Maintenance conditions will engage in Group-Mediated Cognitive Behavioural (GMCB) therapy related to maintaining exercise in their home environment, while women in the Contact conditions will partake in group mediated discussions related to other health issues. The "Forever Free" smoking replase prevention book series (Brandon, Collins, Juliano, & Lazev, 2000) will be distributed to participants in the Relapse Prevention Booklets conditions; however, all groups will receive the same amount of supervised exercise sessions and NRT. Following the termination of the 14 week intervention all participants will be contacted by a trained facilitator, who will deliver 15 minute biweekly (for the first month), monthly (for the next 2 months), and then bimonthly (for last 8 months) intervention strategies over the phone to continue to counsel the women according to her particular group-mediated condition.

Primary end points (i.e., smoking abstinence) will be assessed weekly throughout the 14 week program and through follow-ups at 3, 6, and 12 months. Secondary end points (i.e., fitness, vascular health [e.g., endothelial function, carotid plaque volume], lung function, weight and self-regulatory cognitions) will be assessed at baseline and at week 14 as well as at 12 months. Accelerometers (ACTICALÒ) will be used to obtain an objective measure of physical activity at baseline, week 15 (1 week after the 14 week intervention) and at 6 and 12 months.

The Getting Physical on Cigarettes trial will not only contribute to a better understanding of the role exercise plays as an aid to smoking cessation, but will also explore a means of increasing the cost-effectiveness of long-term smoking cessation programs. The findings resulting from this trial may have important implications for improving the quality of life among individuals who wish to stop smoking, which would, in turn, have a significant impact on the cost of health care to the Canadian public.

ELIGIBILITY:
Participants must meet the following criteria:

* Between the ages of 18 and 65
* Smoking greater than 10 cigarettes per day, have done so for the past 2 years, and want to quit
* Engage in 2 or less 30-minute bouts of moderate or vigorous intensity exercise over the past 6 months
* Absence of any medical condition that is contraindicative for exercise
* not pregnant or intending on being pregnant over the course of the study
* Be able to read and write in English
* Have a telephone or an email account that we can reach you at

Exclusion criteria include:

* Contraindication to regular exercise (e.g., disability, unstable angina)
* Contraindications to using nicotine replacement therapy (NRT)
* Currently exercise more than twice a week for 30 or more minutes each bout at a moderate to vigorous intensity level and have done so for the past 6 months
* On medication for physical and/or mental health reasons that would make compliance with the study protocol difficult or dangerous
* Have substance dependency problems (e.g., alcohol)
* Are pregnant or are planning on becoming pregnant during the next year
* No Medical Doctor approval for exercise or NicoDerm patch (Nicotine Replacement Therapy; NRT)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2009-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Smoking Behaviour | 56 weeks post participant start date
  Continuous smoking behaviour will be measured from week 4-week 14, week26, week 56 (one year following quit). Smoking behaviour will be measured via self-report, breath Carbon Monoxide less than 6 parts per million, saliva cotinine.

SECONDARY OUTCOMES:
Exercise Behaviour | for 56 weeks post participant start
  Exercise behaviour will be measured via Actical accelerometer at baseline, week 14, week 26 and week 56.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D., Principal Investigator — The University of Western Ontario
Locations (1):
- Exercise and Health Psychology Laboratory - The University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Background] Brandon TH, Collins BN, Juliano LM, Lazev AB. Preventing relapse among former smokers: a comparison of minimal interventions through telephone and mail. J Consult Clin Psychol. 2000 Feb;68(1):103-13. doi: 10.1037//0022-006x.68.1.103. PMID 10710845
- [Background] Brandon TH, Meade CD, Herzog TA, Chirikos TN, Webb MS, Cantor AB. Efficacy and cost-effectiveness of a minimal intervention to prevent smoking relapse: dismantling the effects of amount of content versus contact. J Consult Clin Psychol. 2004 Oct;72(5):797-808. doi: 10.1037/0022-006X.72.5.797. PMID 15482038
- [Background] Marcus BH, Albrecht AE, King TK, Parisi AF, Pinto BM, Roberts M, Niaura RS, Abrams DB. The efficacy of exercise as an aid for smoking cessation in women: a randomized controlled trial. Arch Intern Med. 1999 Jun 14;159(11):1229-34. doi: 10.1001/archinte.159.11.1229. PMID 10371231
- [Background] Prapavessis H, Cameron L, Baldi JC, Robinson S, Borrie K, Harper T, Grove JR. The effects of exercise and nicotine replacement therapy on smoking rates in women. Addict Behav. 2007 Jul;32(7):1416-32. doi: 10.1016/j.addbeh.2006.10.005. Epub 2006 Nov 9. PMID 17097814
- [Background] Schnoll RA, Patterson F, Wileyto EP, Tyndale RF, Benowitz N, Lerman C. Nicotine metabolic rate predicts successful smoking cessation with transdermal nicotine: a validation study. Pharmacol Biochem Behav. 2009 Mar;92(1):6-11. doi: 10.1016/j.pbb.2008.10.016. Epub 2008 Oct 31. PMID 19000709
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Prapavessis H, De Jesus S, Fitzgeorge L, Rollo S. Anthropometric and body composition changes in smokers vs abstainers following an exercise-aided pharmacotherapy smoking cessation trial for women. Addict Behav. 2018 Oct;85:125-130. doi: 10.1016/j.addbeh.2018.06.003. Epub 2018 Jun 7. PMID 29902683
- See also: Exercise and Health Psychology Laboratory — http://www.ehpl.uwo.ca